CLINICAL TRIAL: NCT01323829
Title: A Pilot Study: Botulinum Toxin Type A Injections Into Pelvic Muscles for Patients With Refractory High Tone Pelvic Floor Dysfunction
Brief Title: EMG Guided Botulinum Toxin Type A Injections for Refractory High Tone Pelvic Floor Dysfunction
Acronym: BTXA EMG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pelvic and Sexual Health Institute (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Kristene Whitmore, M.D., Medical Director, Pelvic and Sexual Health Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTXA EMG
Record Dates: First submitted 2011-03-24; First posted 2011-03-28 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-05

CONDITIONS: High Tone Pelvic Floor Dysfunction
Keywords: High Tone Pelvic Floor Dysfunction; Botulinum toxin type A; EMG

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: EMG Guidance of Injection — The use of the EMG guidance is the experimental part of the study. We will perform EMG Needle testing in order to pin-point the best location for the patients Botox injections.

SUMMARY:
This is a prospective, pilot, longitudinal study to evaluate the use of EMG guidance for Botox A injection for chronic pelvic pain and HTPFD. The objective of this study is to determine the efficacy of injecting botulinum toxin type A into pelvic floor muscles that are high tone. Patients who have been diagnosed with high tone pelvic floor muscle dysfunction and have failed other treatments will be eligible to participate in this study. Study related procedures will include perineometry readings. Patients will be required to complete 7 questionnaires for this study. These include visual analog scale (scale from 0-10) for pain (VAS), the O'Leary-Sant urinary symptoms and problem questionnaires (ICSI/ICPI), Pelvic Floor Distress Inventory 20 (PFDI-20), the Female Sexual Distress Scale (FSDS), Global Response Assessment Scale and the SF-12 quality of life scale. The use of the EMG guidance is the experimental part of the study. We will perform EMG Needle testing in order to pin-point the best location for the patients Botox injections. This is a prospective, pilot, longitudinal study to evaluate the effect of Botox A injection for chronic pelvic pain and HTPFD.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be diagnosed with High Tone Pelvic Floor Dysfunction(HTPMFD).
* Participant must have tried and failed at least one other conventional mode of therapy for HTPMFD.
* Participant must be a female at least 18 years of age.
* Participant must give written informed consent to participate in this study.
* Participant must be able to make decisions for herself.
* Participant must not be undergoing another procedure at the time of BTX A injection.

Exclusion Criteria:

* Participant is male.
* Patient has a history of past BTX A use
* Patient has had pelvic organ prolapse repair
* Participant is pregnant or intends to get pregnant during the study period or is breastfeeding.
* Participant is unwilling or unable (because of long distance from office) to follow-up.
* Participant has a neuro-modulator device implanted.
* Participant has a known bleeding disorder or is on anticoagulation.
* Participant has a known hypersensitivity to BTX A.
* Participant has a pre-existing neuromuscular disorder such as amytrophic lateral sclerosis, motor neuropathy, myasthenia gravis or Lambert-Eaton syndrome.
* Participant with skin infection at the perineum at the site of injection.

Ages: 18 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-11; Primary Completion 2013-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the use of EMG guidance for Botox A injection for chronic pelvic pain and HTPFD. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kristene E Whitmore, MD, Principal Investigator — Pelvic and Sexual Health Institute
Locations (1):
- Pelvic and Sexual Health Institute, Philadelphia, Pennsylvania, United States